CLINICAL TRIAL: NCT00132028
Title: A Phase II Trial of Suberoylanilide Hydroxamic Acid (NSC-701852) for Recurrent or Primary Refractory Hodgkin's Lymphoma
Brief Title: Vorinostat in Treating Patients With Relapsed or Refractory Advanced Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03071; NCI-2012-03071 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA032102 (NIH); S0517 (Other: SWOG); S0517 (Other: CTEP)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2013-01

CONDITIONS: Adult Favorable Prognosis Hodgkin Lymphoma; Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Lymphocyte Predominant Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nodular Lymphocyte Predominant Hodgkin Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Adult Unfavorable Prognosis Hodgkin Lymphoma; Recurrent Adult Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Vorinostat

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive oral vorinostat twice daily on days 1-14. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses of therapy beyond CR.
  Interventions: Drug: vorinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well vorinostat works in treating patients with relapsed or refractory advanced Hodgkin's lymphoma. Vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response probability (complete, complete unconfirmed, and partial) in patients with relapsed or refractory Hodgkin's lymphoma.

II. To estimate 1-year progression-free survival and overall survival in patients with relapsed or refractory Hodgkin's lymphoma treated with SAHA.

III. To assess the toxicity profile of SAHA in this patient population. IV. To perform gene expression profiling on tumor tissue before and after treatment in order to explore in a preliminary manner the association between response and specific gene expression results.

OUTLINE: This is a multicenter study.

Patients receive oral vorinostat twice daily on days 1-14. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses of therapy beyond CR.

After completion of study treatment, patients are followed every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed relapsed/refractory Hodgkin's lymphoma of any subtype; patients with lymphocyte predominant Hodgkin's disease (LPHD) are also eligible; clear evidence of disease progression or lack of response after the most recent therapy, including local radiation is required
* Patients must be willing to submit specimens for correlative studies
* All patients must have bidimensionally measurable disease documented within 28 days prior to registration; patients with non-measurable disease in addition to measurable disease must have all non-measurable disease assessed within 42 days prior to registration
* Patients must have unilateral bone marrow aspirate and biopsy performed within 42 days prior to registration
* Patients may have had up to five prior chemotherapy regimens
* Patients must have completed chemotherapy at least 28 days prior to registration and all toxicities must have resolved (in the opinion of the treating investigator); if last regimen included nitrosoureas or mitomycin then 42 days must have elapsed since completion of treatment; patients must not have taken valproic acid, or another histone deacetylase inhibitor, for at least 14 days prior to registration
* Patients must have completed all radiotherapy at least 14 days prior to registration and all toxicities must have resolved (in the opinion of the treating investigator)
* Patients who relapse after autologous stem cell transplant may be enrolled if they are at least three months after transplant, and after allogeneic transplant if they are at least one year posttransplant; patients should have no active related infections (i.e., fungal or viral); in the case of allogeneic transplant relapse, there should be no active acute graft versus host disease (GvHD) of any grade, and no chronic graft versus host disease other than mild skin, oral, or ocular GvHD not requiring systemic immunosuppression
* Patients must have a Zubrod performance status of 0-2
* Patients must have a CT scan of the chest/abdomen and pelvis performed within 28 days prior to registration
* Patients must not have clinical evidence of central nervous system involvement by lymphoma; any laboratory or radiographic tests performed to assess CNS involvement must be negative within 42 days of registration
* Serum LDH must be measured within 28 days prior to registration
* Absolute neutrophil count >- 1,000/mcL
* Platelet count >= 100,000/mcL
* SGOT/SGPT < 2.5 x the institutional upper limit of normal
* Serum creatinine < 2 x the institutional upper limit of normal
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biological composition to SAHA are ineligible
* Patients must not have plans to receive concurrent hormonal, biological or radiation therapy; patients with potentially curative options such as salvage therapy with chemotherapy or hematopoietic stem cell transplant (HSCT) are not eligible
* Patients with a history of prior myocardial infarction, unstable angina, or stroke within 6 months are ineligible
* Patients known to be HIV-positive and receiving combination antiretroviral therapy are ineligible; in addition, HIV-positive patients not receiving combination antiretroviral therapy are also ineligible
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer for which the patient has been disease-free for five years
* Pregnant or nursing women may not participate; women or men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kirschbaum, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group (SWOG) Research Base, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SAHA (Vorinostat): Patients receive vorinostat 400 mg/day on days 1-14 of every 21-day cycle. Patients continue treatment until progression.
Period: Overall Study
Arm/Group | SAHA (Vorinostat)
Started | 27
Eligible | 25
Eligible and Began Protocol Therapy | 25
Completed | 0 (Since there was no maximum number of cycles, patients could not "complete" treatment.)
Not Completed | 27
Not completed — Adverse Event | 7
Not completed — Death | 2
Not completed — Lack of Efficacy | 11
Not completed — Withdrawal by Subject | 2
Not completed — not eligible | 2
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | SAHA (Vorinostat)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 41.6 [19.9 to 71.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Assess Number of Patients Who Achieve Confirmed and Unconfirmed Complete Response (CR) or Partial Response (PR)
Description: Complete Response(CR) is a complete disappearance of all disease with the exception of nodes. No new lesions. previously enlarged organs must have regressed and not be palpable. Bone marrow(BM) must be negative if positive at baseline. Normalization of markers. CR Unconfirmed (CRU) does not qualify for CR above, due to a residual nodal mass or an indeterminate BM. Partial Response(PR) is a 50% decrease in the SPD for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes.
Time Frame: after every 3 cycles on treatment
Population: All patients who started treatment were included in assessing response estimates.
Measure: Number; unit: participants
Arm/Group | SAHA (Vorinostat)
Number analyzed (Participants) | 25
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 1
  Unconfirmed Complete Response (UCR) | 0
  Unconfirmed Partial Response (UPR) | 0
  No Response | 24

2. Secondary Outcome: Progression-Free Survival
Description: Measured from date of registration to date of first observation of progression or death, or last contact date. Progression is defined as a 50% increase in sum of products of greatest diameters (SPD) of target measurable lesions over the smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline; appearance of a new lesion/site; unequivocal progression of non-measurable disease in the opinion of the treating physician; death due to disease without prior documentation of progression.
Time Frame: after every 3 cycles on treatment, then every 6 months for 2 years, then annually for a total of 5 years.
Population: All eligible patients who started treatment were included in assessing progression-free survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SAHA (Vorinostat)
Number analyzed (Participants) | 25
months | 4.8 [3.4 to 13.2]

3. Secondary Outcome: Overall Survival
Description: Measured from date of registration to death, or last contact date
Time Frame: after every 3 cycles on treatment, then every 6 months for 2 years, then annually for a total of 5 years.
Population: All eligible patients who started treatment were included in assessing overall survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SAHA (Vorinostat)
Number analyzed (Participants) | 25
months | 15.7 [6.6 to 34.1]

ADVERSE EVENTS:
Time Frame: After every 21-day cycle while on protocol treatment
Arm/Group | SAHA (Vorinostat)
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SAHA (Vorinostat) (N=25)
Hemoglobin (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 1
Creatinine (Investigations) | 1
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1
Platelets (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAHA (Vorinostat) (N=25)
Hemoglobin (Blood and lymphatic system disorders) | 20
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 16
Pain - Stomach (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 8
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 4
Flu-like syndrome (General disorders) | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 2
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 7
Alkaline phosphatase (Investigations) | 7
Bilirubin (hyperbilirubinemia) (Investigations) | 2
Creatinine (Investigations) | 6
Leukocytes (total WBC) (Investigations) | 7
Lymphopenia (Investigations) | 11
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4
Platelets (Investigations) | 11
Weight loss (Investigations) | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 10
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 3
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 3
Pain - Head/headache (Nervous system disorders) | 5
Taste alteration (dysgeusia) (Nervous system disorders) | 2
Proteinuria (Renal and urinary disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less